CLINICAL TRIAL: NCT04488328
Title: Effect of Magnetic Therapy and Moderate Aerobic Exercise on Post Thyroidectomy Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Eid, assistant professor of physical therapy for surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 68m
Record Dates: First submitted 2020-07-17; First posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Magnetic Therapy Group (Experimental): patients received the routine medical treatment (Bisphosphonates, Calcium, and Vitamin D) in addition to pulsed magnetic therapy on the pelvic region for 12 weeks
  Interventions: Other: patients received the routine medical treatment in addition to pulsed magnetic therapy and moderate-intensity aerobic exercise for 12 weeks
- Exercise group (Experimental): patients received the routine medical treatment in addition to moderate-intensity aerobic exercise for 12 weeks
  Interventions: Other: patients received the routine medical treatment in addition to pulsed magnetic therapy and moderate-intensity aerobic exercise for 12 weeks
- Combined Magnetic Therapy and Exercise Therapy group (Experimental): patients received the routine medical treatment in addition to pulsed magnetic therapy and moderate-intensity aerobic exercise for 12 weeks
  Interventions: Other: patients received the routine medical treatment in addition to pulsed magnetic therapy and moderate-intensity aerobic exercise for 12 weeks

INTERVENTIONS:
Other: patients received the routine medical treatment in addition to pulsed magnetic therapy and moderate-intensity aerobic exercise for 12 weeks — patients received the routine medical treatment in addition to pulsed magnetic therapy and moderate-intensity aerobic exercise for 12 weeks(3 sessions/ week)

SUMMARY:
Objectives; This study was conducted to investigate the effect of pulsed magnetic therapy and aerobic exercise on post thyroidectomy osteoporosis.

Methods; Forty-five female patients, age ranged from 40 to 50 years old with osteoporotic changes in hip and pelvic region post thyroidectomy, were included in this study. They were selected from Endocrinology private clinics. They were assigned randomly into three groups, equal in number. Magnetic Therapy Group (group A); patients received the routine medical treatment (Bisphosphonates, Calcium, and Vitamin D) in addition to pulsed magnetic therapy on the pelvic region for 12 weeks (3 sessions/ week). Exercise group(group B); patients received the routine medical treatment in addition to moderate-intensity aerobic exercise for 12 weeks (3 sessions/week). Combined Magnetic Therapy and Exercise Therapy group (group C): patients received the routine medical treatment in addition to pulsed magnetic therapy and moderate-intensity aerobic exercise for 12 weeks. Evaluation of the three groups was performed at baseline and after 12 weeks of treatment by dual energy x-ray absorptiometry (DEXA).

ELIGIBILITY:
Inclusion Criteria:

* All participants had undergone thyroidectomy since 6 months and had cognitive and educational level enough to understand the requirements of the study

Exclusion Criteria:

* All Patients with malignancies or receiving radiotherapy or chemotherapy, skin diseases, deep venous thrombosis or venous insufficiency, sensory impairment, renal failure, recent therapy with immunosuppressant or anticonvulsants, psychological problems or alcoholic drinkers were excluded from this study.

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Osteoporosis changes | 12 weeks
  BMD by DEXA on each group

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Eid, Principal Investigator — Cairo University
Locations (1):
- Marwa Eid, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided